CLINICAL TRIAL: NCT05207306
Title: Postoperative Analgesic Effect of Ultrasound-guided Thoracoabdominal Nerves Block Through Perichondrial Approach in Patients Undergoing Laparoscopic Cholecyctectomy: A Randomized Controlled Study
Brief Title: Comparision of M-TAPA Versus TAPB After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, Assistant clinical professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2111-040-1270
Record Dates: First submitted 2022-01-02; First posted 2022-01-26 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain, Acute
Keywords: cholecystectomy; thoracoabdominal nerves block; transversus abdominis plane block; interfascial plane block; regional analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A prospective randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded to the allocation, because that investigator performed nerve block after induction of anesthesia. The outcome assessor not involved in this study will investigate the outcomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) group (Experimental): Patients receiving right M-TAPA.
  Interventions: Procedure: Type of interfascial plane block
- Subcostal transversus abdominis plane block (subcostal TAPB) group (Experimental): Patients receiving right subcostal TAPB.
  Interventions: Procedure: Type of interfascial plane block

INTERVENTIONS:
Procedure: Type of interfascial plane block — In the M-TAPA group, after finding the right 10th costal cartilage using ultrasound guidance, a anesthesiologist inject 0.375% ropivacaine 15ml into the lower aspect of the chondrium. Perform left M-TAPA in the same way.
  In the subcostal TAPB group, a anesthesiologist inject 0.375% ropivacaine 15ml into end of right rectus abdominis muscle using ultrasound guidance. Perform left subcostal TAPB in the same way.

SUMMARY:
This randomized controlled study is designed to evaluate the postoperative analgesic effect of the ultrasound-guided modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) in patients undergoing laparoscopic cholecystectomy. The investigators hypothesized that the US-guided M-TAPA would be more effective in postoperative pain control than the US-guided subcostal transversus abdominis plane block (TAPB).

DETAILED DESCRIPTION:
Patients (Age>18 years) undergoing elective laparoscopic cholecystectomy are randomly allocated to receive bilateral US-guided M-TAPA (n=30) or bilateral subcostal TAPB (n=30) using 0.375% ropivacaine 15ml (total 30ml) before surgical incision. The blinded investigator evaluates each patient's parameters (Numeric rating scale, nausea, vomiting, pruritis, and patient satisfaction) at 1, 2, 4, 6, 12hours postoperatively, and immediately before discharge. The primary outcome is pain severity evaluated by a NRS at 12hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective laparoscopic cholecystectomy
* American Society of Anesthesiologists (ASA) physical classification I-II

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical classification III or more
* Chronic pain, chronic analgesic or antidepressant or anticonvulsant use
* Allergies to anesthetic or analgesic medications used in the protocol
* Single port laparoscopic cholecystectomy
* Patients with infection at the abdominal wall
* Medical or psychological disease that can affect the treatment response
* Do not understand our study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Maximum postoperative pain score during 12hours postoperatively | at 12hour postoperatively.
  maximum pain score measured by the 11-pointed numeric rating scale (0: none/10: worst pain) during 12hours postoperatively

SECONDARY OUTCOMES:
Postoperative pain score at rest | at 1, 2, 4, 6, 12hours postoperatively, and immediately before discharge
  Change in the pain severity measured by the 11-pointed numeric rating scale (0: none/10: worst pain) pain score at resting
Postoperative pain score during coughing | at 1, 2, 4, 6, 12hours postoperatively, and immediately before discharge
  Change in the pain severity measured by the 11-pointed numeric rating scale (0: none/10: worst pain) pain score during coughing
Patient satisfaction before discharge | at immediately before discharge
  Patient satisfaction measured by the 7-pointed Likert scale. (1: Strongly dissatisfaction/ 7: Strongly satisfaction)
Occurrence rate of postoperative nausea, vomiting | at 1, 2, 4, 6, 12hours postoperatively, and immediately before discharge.
  Incidence of postoperative nausea and vomiting (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Please Select An Option, South Korea

REFERENCES:
- [Background] Aikawa K, Tanaka N, Morimoto Y. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides a sufficient postoperative analgesia for laparoscopic sleeve gastrectomy. J Clin Anesth. 2020 Feb;59:44-45. doi: 10.1016/j.jclinane.2019.06.020. Epub 2019 Jun 15. No abstract available. PMID 31212124
- [Background] Ueshima H, Hiroshi O. RETRACTED: Thoracoabdominal nerves block through the perichondral approach for effective perioperative analgesia during upper abdominal surgery. J Clin Anesth. 2020 Feb;59:7. doi: 10.1016/j.jclinane.2019.06.008. Epub 2019 Jun 5. No abstract available. PMID 31176261 (Retraction: PMID 35551833 J Clin Anesth. 2022 Sep;80:110839)
- [Background] Taylor R Jr, Pergolizzi JV, Sinclair A, Raffa RB, Aldington D, Plavin S, Apfel CC. Transversus abdominis block: clinical uses, side effects, and future perspectives. Pain Pract. 2013 Apr;13(4):332-44. doi: 10.1111/j.1533-2500.2012.00595.x. Epub 2013 Feb 13. PMID 22967210
- [Background] Oksar M, Koyuncu O, Turhanoglu S, Temiz M, Oran MC. Transversus abdominis plane block as a component of multimodal analgesia for laparoscopic cholecystectomy. J Clin Anesth. 2016 Nov;34:72-8. doi: 10.1016/j.jclinane.2016.03.033. Epub 2016 May 2. PMID 27687350
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Turan M, Gumus Demirbilek S. Comparison of the effects of modified pectoral nerve block and erector spinae plane block on postoperative opioid consumption and pain scores of patients after radical mastectomy surgery: A prospective, randomized, controlled trial. J Clin Anesth. 2019 May;54:61-65. doi: 10.1016/j.jclinane.2018.10.040. Epub 2018 Nov 3. PMID 30396100